CLINICAL TRIAL: NCT00588497
Title: Characterization of the Essure System Tubal Sterilization Using Ultrasound and X-Ray
Status: Completed | Type: Observational
Sponsor: Mayo Clinic (Other)
Responsible Party: Abimbola O. Famuyide, M.D., Chair, Division of Gynecology, Mayo Clinic, Rochester, MN
Other Study IDs: 628-04
Record Dates: First submitted 2007-12-22; First posted 2008-01-08 (Estimated); Last update posted 2011-05-23 (Estimated); Status verified 2011-05

CONDITIONS: Tubal Sterilization
Keywords: female sterilization, micro-insert, hysteroscopy

STUDY DESIGN:
Time Perspective: Prospective

GROUPS / COHORTS (1):
- Study Group: Twenty-five subjects for this study will be recruited from patients who have requested a form of permanent sterilization, and who, after considering all the options, choose the trans-cervical hysteroscopic sterilization for this end. Any subject who is deemed suitable for the micro-insert hysteroscopic sterilization system (Essure micro-insert system, Conceptus Incorporated, Mountain View, California) placement will be offered the opportunity to participate in the study.
  Interventions: Procedure: Micro-insert hysteroscopic sterilization; Radiation: Plain abdominal Xray; Procedure: Pelvic Ultrasound; Radiation: Hysterosalpingogram

INTERVENTIONS:
Procedure: Micro-insert hysteroscopic sterilization — Placement of micro-inserts transcervically with the aid of a hysteroscope
Radiation: Plain abdominal Xray — Performed immediately after micro-inserts placement and at 3 months
Procedure: Pelvic Ultrasound — Performed immediately after micro-inserts placement and at 3 months.
Radiation: Hysterosalpingogram — Performed 3 months after micro-inserts placement

SUMMARY:
Tubal sterilization is the most prevalent form of contraception in the United States and the world. Currently, approximately half of these are performed with a laparoscope and half through a mini-laparotomy after delivery. Micro-insert hysteroscopic sterilization system received FDA approval for elective sterilization in 2003. Compared to other forms of female sterilization, this procedure is minimally invasive and does not require entering the abdominal cavity. In addition, it is at least as effective in preventing pregnancy as other forms of tubal occlusion. Given the distinct advantages of this method, it could become the preferred method of tubal sterilization for physicians and their patients. Currently, there is no published data concerning the appearance of the micro-inserts system using other imaging modalities that are commonly used in gynecologic practice. As the use of this device becomes more widespread it will be more commonly encountered in radiographic imaging performed as part of routine patient care. The main objective of this study is to provide important descriptive data concerning the ultrasonographic and x-ray appearance of the micro-insert hysteroscopic sterilization device. An additional objective of this study is to identify characteristics on plain film and ultrasound (US) that correlate with tubal occlusion or patency.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients requesting sterilization

Exclusion Criteria:

* Unsuccessful placement of the hysteroscopic sterilization system in one or both fallopian tubes. In addition, a patient will not be offered the opportunity to participate in the study if there are any conditions that would preclude attempted placement of the hysteroscopic sterilization system. These include hypersensitivity to nickel-titanium or contrast media, current or recent pregnancy (within the previous six weeks), active genital tract infection, prior tubal ligation, or known congenital uterine malformation.

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Twenty-five subjects for this study will be recruited from patients who have requested a form of permanent sterilization, and who, after considering all the options, choose the trans-cervical hysteroscopic sterilization for this end. Any subject who is deemed suitable for the micro-insert hysteroscopic sterilization system (Essure micro-insert system, Conceptus Incorporated, Mountain View, California) placement will be offered the opportunity to participate in the study. Consent will be documented on a Mayo Clinic patient consent form at the time the decision is made to schedule the procedure.
Sampling Method: Non-Probability Sample
Enrollment: 25 (Actual)
Dates: Start 2004-02; Primary Completion 2006-03 (Actual); Study Completion 2006-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Abimbola O. Famuyide, M.D., Principal Investigator — Mayo Clinic, Rochester, MN
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States